CLINICAL TRIAL: NCT07170826
Title: Evaluation of a Therapeutic Education Program on Self-image in Patients With Chronic Inflammatory Rheumatic Diseases
Acronym: IMAG'RIC
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250978; IDRCB (Other: 2025-A01584-45)
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Chronic Inflammatory Rheumatic Diseases
Keywords: Chronic Inflammatory Rheumatic diseases; Therapeutic patient education
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self questionnaire — Rosenberg Scale, SF36, MBRSQ
Other: interview — Semi-structured individual interviews

SUMMARY:
Chronic inflammatory rheumatic diseases (CIRD), like all chronic somatic disease, can impair self-esteem and self-image in affected individuals. Numerous studies conducted in this population have confirmed this fact. Therapeutic patient education (TPE) programs aim to help patients acquire self-care and adaptive skills. However, there is a near-total absence of workshops specifically dedicated to self-image in TPE programs for CIRD. Such educational interventions have shown their effectiveness in contexts such as cancer and obesity. Our study aims to evaluate their effectiveness for patients with CIR.

DETAILED DESCRIPTION:
A chronic disease is a long-term, progressive illness that affects the daily life of the person affected. The onset of the disease is a major upheaval, a moment of rupture between a before and an after. Physical functions and appearance can be altered by the disease (deformities, stiffness… in the case of rheumatic diseases) and by treatments.

According to Schilder, body image is "the way our body appears to ourselves." It can be defined as the set of perceptions, emotions, and thoughts related to appearance. It consists of perceptions but also of representations and feelings, which are built and evolve throughout the individual's experience. It is not limited to physical appearance and properties. It is the foundation of identity.

The disease affects the body, but also has an impact on self-perception, self-esteem, and even identity.

The literature highlights the importance of using qualitative research in addition to quantitative methods to grasp the full complexity of body image.

Despite the progress and effectiveness of treatments, recent studies showed that patients with chronic inflammatory rheumatic diseases (CIRD) have an unsatisfactory, disturbed body image. Literature data also reveal that self-esteem and quality of life in this population are lower than in the general population.

Most studies focused on the consequences of the disease, and very few on the actions taken to address these difficulties encountered by patients, even though such actions are recommended.

Therapeutic patient education (TPE) is support offered to the patient and their relatives so they can take ownership of their disease. TPE is a comprehensive approach that meets the patient's needs and aims to maintain and/or improve quality of life with the illness.

Most therapeutic education workshops related to self-image are proposed in the context of cancer, psychiatric disorders, or obesity. Body image is rarely the direct subject of a workshop in programs aimed at patients with CIRD.

A few studies on the impact of image consulting workshops have been conducted in oncology, but very few in the context of other diseases, including rheumatic conditions. Existing studies show an improvement in self-image, self-esteem, and quality of life after educational interventions, thus a real benefit for patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Suffering from chronic inflammatory rheumatism (rheumatoid arthritis, spondyloarthritis, psoriatic arthritis)
* Having agreed to follow the therapeutic education programme offered by the department as part of routine care
* Not opposed to participating in the research

Exclusion Criteria:

* People who do not speak or read French
* Current pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will consist of patients with RIC (rheumatoid arthritis, spondyloarthritis, psoriatic arthritis) participating in the ETP programme
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate a therapeutic patient education intervention focused on self-image in patients with chronic inflammatory rheumatic diseases | 3 months following completion of the 'self-image' module
  Multidimensional Body-Self Relations Questionnaire (MBSRQ)

SECONDARY OUTCOMES:
To evaluate a therapeutic patient education intervention on each domain of self-image | 3 months following completion of the 'self-image' module
  Measurement of each subscale of the Multidimensional Body-Self Relations Questionnaire (MBSRQ)
To evaluate a therapeutic patient education intervention focused on self-image in relation to self-esteem. | 3 months following completion of the 'self-image' module
  Rosenberg Self-Esteem Scale before participation : min = 10, max=40
To evaluate a therapeutic patient education intervention focused on self-image in relation to quality of life. | 3 months following completion of the 'self-image' module
  Measurement of the quality of life score using the SF-36 questionnaire
To explore body image in patients after participating in therapeutic education workshops on self-image. | 4 months following completion of the 'self-image' module
  Data from individual qualitative interviews (inductive approach).

CONTACTS AND LOCATIONS:
Overall Officials: Marie Laure TOURNEUR, Marie Laure, Principal Investigator — AP-HP - Hôpital Cochin - Service de rhumatologie.
Locations (1):
- Hôpital Cochin - Service de rhumatologie -27 rue du Faubourg St Jacques, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No